CLINICAL TRIAL: NCT01588743
Title: Effects of Short-term Intensive Insulin Therapy on Insulin Resistance and Insulin Secretion in Newly Diagnosed Lean and Obese Type 2 Diabetes Patients
Brief Title: Effects of Short-term Intensive Insulin Therapy in Newly Diagnosed Type 2 Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Li Guangwei (Other)
Responsible Party: Sponsor-Investigator, Li Guangwei, Professor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prof. Li Guangwei
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

INTERVENTIONS:
Drug: insulin aspart — Insulin Aspart will be administrated by insulin pump with an initial dose of 0.4-0.6u/kg body weight, of which 50% basal rate and the other 50% bolus dose. Time interval for administration will be as follows: 0-3Am-9Am-12Am-5Pm-9Pm-0Am. Specific adjustment will be made according to individual difference.

SUMMARY:
It is well known that Long-term hyperglycemia (also known as glucose toxicity) contribute to impairment in islet β-cell function and development of insulin resistance. A growing body of evidence also indicates that this impairment inβ-cell function and insulin action could be restored after hyperglycemia is corrected by short-term intensive insulin therapy. In this study, we are determined to use the golden standard of insulin sensitivity evaluation in vivo-hyperinsulinemia euglycemic glucose clamp-to estimate insulin resistance improvement in patients before and after intensive insulin therapy, investigate first phase insulin secretion to evaluate β-cell function, examine the changes in insulin resistance and insulin secretion resulting from normalization of plasma glucose levels in both lean and obese patients by insulin pump therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 to 60 years old
* Duration of diabetes: newly diagnosed type 2 diabetes (duration of diabetes less than 1 year) and haven't taken any antidiabetic medication.
* Fasting blood glucose is above 11.0mmol/L.
* Half of the patients with BMI below 24 and the other half with BMI above 24.

Exclusion Criteria:

* type 1 diabetes mellitus
* type 2 diabetes patients with intercurrent illness (ketoacidosis, infection or any other acute stress)
* Presence of auto-immune disease, hepatic or renal disease or any concomitant disease is not allowed.
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 12 months.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
AUC75-120 of Glucose Infusion Rate (GIR) | after 2 weeks insulin pump intensive therapy, and one-year follow-up after termination of treatments

SECONDARY OUTCOMES:
AUC0-10 of Acute Insulin Response (AIR) during IVGTT | after 2 weeks insulin pump intensive therapy, and one-year follow-up after termination of treatments

CONTACTS AND LOCATIONS:
Overall Officials: Guangwei Li, Principal Investigator — China-Japan Friendship Hospital

REFERENCES:
- [Derived] Wang H, Kuang J, Xu M, Gao Z, Li Q, Liu S, Zhang F, Yu Y, Liang Z, Zhao W, Yang G, Li L, Wang Y, Li G. Predictors of Long-Term Glycemic Remission After 2-Week Intensive Insulin Treatment in Newly Diagnosed Type 2 Diabetes. J Clin Endocrinol Metab. 2019 Jun 1;104(6):2153-2162. doi: 10.1210/jc.2018-01468. PMID 30629195